CLINICAL TRIAL: NCT01528189
Title: Effect of Hyperinsulinemic Normoglycemic Clamp (HINC) on Infectious Complications Following Major Abdominal Surgery. A Randomized Controlled Trial.
Brief Title: Effect of High Dose Insulin on Infectious Complications Following Major Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ralph Lattermann, Assistant Professor, Department of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-01
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2024-06

CONDITIONS: Surgical Site Infection After Major Surgery
Keywords: Insulin, surgery, infection
MeSH Terms: conditions — Insulin Resistance; Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard glucose management (Placebo Comparator): Arterial-blood glucose levels will be checked at induction of anesthesia and every 30 - 60 min thereafter with an StatStrip Xpress® (Nova Biomedical, MA, USA) ( A blood glucose level above 10 mmol/l will be treated with a 2U bolus of IV insulin (Humulin® R regular insulin, Eli Lilly and Company, Indianapolis, IN) followed by a 1 U/hour drip infusion adjusted according to a standard sliding scale
  Interventions: Other: Standard glucose management
- Hyperinsulinemic normoglycemic clamp (Active Comparator): The blood glucose level will be checked prior to intubation. A 2U bolus of IV insulin will be given if blood glucose level is higher than 6 mmol/l, followed by an IV infusion of 2 U/kg/min (0.12 U/kg/hour). Dextrose 20% (D20W®) will be titrated to maintain blood glucose between 4 and 6 mmol/l. Blood glucose levels will be measured at 5-30 min intervals with a to ensure normoglycemia. At the end of surgery, the insulin infusion will be stopped, and the dextrose infusion weaned off in the post anesthesia care unit.
  Interventions: Other: Hyperinsulinemic normoglycemic clamp

INTERVENTIONS:
Other: Hyperinsulinemic normoglycemic clamp — Patients will receive an IV infusion of 2 mU/kg/min (0.12 U/kg/hour) starting in the operating room. Dextrose 20% will be titrated to maintain blood glucose between 4 and 6 mmol/l. At the end of surgery, the insulin infusion will be stopped and the dextrose infusion weaned off in the postanesthesia care unit.
  Arms: Hyperinsulinemic normoglycemic clamp
Other: Standard glucose management — Blood glucose levels will be treated by a standard insulin sliding scale.
  Arms: Standard glucose management

SUMMARY:
Despite improvements in surgical techniques and perioperative care, the high incidence of postoperative surgical site infections remains a major problem in patients undergoing major abdominal surgery (liver, pancreatic and colorectal surgery).

Using the hyperinsulinemic-normoglycemic clamp technique, i.e. continuous infusion of insulin combined with dextrose titrated to "clamp" blood glucose between 4 and 6 mmol/L, we successfully established and preserved normoglycemia during the perioperative period. Our objective of this study is to determine if the maintenance of perioperative normoglycemia by a hyperinsulinemic normoglycemic clamp reduces the rates of incisional and space/ surgical site infections following abdominal surgery (liver, pancreatic and colorectal surgery).

DETAILED DESCRIPTION:
This randomized, open-label, controlled trial will be performed in adult (>18 years old) patients scheduled for elective open abdominal aortic aneurysm repairs and open hepatobiliary procedures including liver resections, pancreatectomies, duodenectomies, gastrojejunostomies, choledochojejunostomies and hepaticojejunostomies) at the Royal Victoria Hospital (RVH), McGill University Health Centre (MUHC), Montreal, QC, Canada.

Inclusion criteria: above 18 years old, scheduled for elective open abdominal aortic aneurysm repairs and open hepatobiliary procedures.

Exclusion criteria: inability to give consent, current wound infection, previous surgery at the same site within the preceding 30 days, allergy to insulin.

RECRUITMENT

Initial contact prior to surgery will be made by a research team member not involved in the care of the patient who will explain the research project and obtain written consent.

Consenting patients will then be randomized with the assistance of a computerized randomization system.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* elective liver, pancreatic or colorectal surgery
* ability to give informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | for 30 days after surgery
  Surgical site infections will be defined according to the CDC's NNIS system.

SECONDARY OUTCOMES:
Surgical morbidity | 30 days after surgery
  Surgical morbidity in the 30 days following the operation will be assessed as per Clavien score.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Lattermann, MD PhD, Principal Investigator — Department of Anaesthesia, McGill University Health Center
Locations (3):
- Canada (2):
  - Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- Hospital Clinico Universidad de Chile, Independencia, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Omiya K, Nakadate Y, Sato H, Koo BW, Schricker T. Accuracy of the Nova StatStrip(R) glucometer in patients undergoing major abdominal surgery: an observational study. Can J Anaesth. 2023 Dec;70(12):1970-1977. doi: 10.1007/s12630-023-02606-z. Epub 2023 Nov 2. PMID 37919630
- [Derived] Omiya K, Sato H, Sato T, Nooh A, Koo BW, Kandelman S, Schricker T. The Quality of Preoperative Glycemic Control Predicts Insulin Sensitivity During Major Upper Abdominal Surgery: A Case-Control Study. Ann Surg Open. 2023 Jan 12;4(1):e234. doi: 10.1097/AS9.0000000000000234. eCollection 2023 Mar. PMID 37600876
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Omiya K, Koo BW, Sato H, Sato T, Kandelman S, Nooh A, Schricker T. Randomized controlled trial of the effect of hyperinsulinemic normoglycemia during liver resection on postoperative hepatic function and surgical site infection. Ann Transl Med. 2023 Mar 15;11(5):205. doi: 10.21037/atm-22-3721. PMID 37007572